CLINICAL TRIAL: NCT00776607
Title: Randomized, Controlled, Parallel-Group Prospective Study to Investigate the Clinical Effectiveness of Early Insulin Treatment in Patients With Latent Autoimmune Diabetes in Adults
Brief Title: Randomized Controlled Trial of Insulin Versus Tablets for Latent Autoimmune Diabetes in Adults (LADA)
Acronym: LIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abertawe Bro Morgannwg University NHS Trust (Other Government)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Dr Sinead Brophy, Swansea University.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-004662-14; ISRCTN63815121; 07/MRE09/8
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-09

CONDITIONS: Latent Autoimmune Diabetes in Adults LADA
Keywords: LADA; Latent autoimmune diabetes in adults; Type 1.5; Slowly progressive type 1 diabetes
MeSH Terms: conditions — Latent Autoimmune Diabetes in Adults | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin (Experimental): Insulin: NovoMix 30. Patients will be given advice on diet and exercise and life style and will be started on NovoMix 30, one dose of 6 U at the evening/main meal.
  Interventions: Drug: NovoMix 30
- Tablet (Active Comparator): Patients will progress from lifestyle modification to metformin, to metformin with Rosiglitazone and finally insulin depending on HbA1c levels.
  Interventions: Drug: Tablet treatment

INTERVENTIONS:
Drug: NovoMix 30 — Insulin arm: Patients will be given advice on diet and exercise and life style and will be started on NovoMix 30, one dose of 6 U at the evening/main meal. Dose will be adjusted in increments of 2-6U depending on fasting glucose level When total dose equals 16 U patient will be started on 4 units with breakfast and continue with 16 units with evening meal. Breakfast and/or evening meal dose will be adjusted where necessary at increments of 2-6 U depending on fasting and/or pre-evening meal glucose level. Patient needs to keep a daily diary of insulin doses taken.
  Arms: Insulin
Drug: Tablet treatment — Step 1: Lifestyle modification. If HbA1c at 7%+ or if on metformin/sulphonylurea go to step 2. Step 2: Glucophage. If HbA1c of 7%-7.5% give 500mg x 1 per day. If HbA1c 7.6%-8.0%, week 1 - 500mg x 1 day and then 500mg x 2 day. If HbA1c 8.0%+ then 500mg x 3 per day (Titrated). If HbA1c remains 7%+ give additional tablet until 2gms per day then progress to Step 3. Step 3: Rosiglitazone. HbA1c of 7%+ give 4 mg per day. If HbA1c remains 7%+ titrate to maximal dose 4 mg twice daily +/-Metformin. If HbA1c remains 7% + for an 3 months move to step 4. Before initiation of Rosiglitazone repeat medical history with special emphasis on cardiovascular disease, if patient has a history of CVD move to Step 4 (insulin). Any adverse events suggestive of heart disease move to step 4. Step 4: Insulin (oral agents will be stopped). Initiation of insulin will the same as for the insulin arm and will follow the protocol detailed in the Insulin arm.
  Arms: Tablet

SUMMARY:
Background: Latent autoimmune diabetes in adults [LADA] is a type 1 diabetes that is slowly developing. This means many people are treated as having type 2 diabetes at diagnosis as they are adults who are not immediately insulin dependent. LADA can be distinguished from type 2 diabetes by antibody tests. Patients who are antibody positive have an autoimmune reaction which is similar to that of type 1 diabetes and is not found in type 2 diabetes. We would like to examine the best way of treating LADA in the early phase of the conditions, with tablets (similar to type 2 diabetes) or with insulin (similar to type 1 diabetes).

Methods/Design: This is an open parallel group prospective randomised trial. Participants need to have a GAD antibody test results of 101 WHO units or more and a diagnosis of diabetes not requiring insulin at diagnosis. Participants will need to have been diagnosed within 12 months and not treated with insulin at study entry. They will be randomised to receive either insulin (NovoMix 30) or tablets (diet treated followed by metformin followed by glitazone (with or without metformin) followed by insulin). Primary outcome assessment will be for change in HbA1c and change in fasting C-peptide over 24 months. Secondary outcome measures will include Quality of life, GAD antibody levels, adverse events, inflammatory markers, insulin resistance, and markers of the metabolic syndrome.

Discussion: This study seeks the best treatment for early LADA in terms of maintaining glycaemic control and maintaining natural insulin production.

ELIGIBILITY:
Inclusion Criteria:

1. Male, non-fertile female (i.e., post menopausal, post hysterectomy, or sterilized by tubal ligation) or female of childbearing potential using a medically approved birth control method.
2. The patient has a diagnosis of diabetes mellitus according to WHO classification.
3. The patient has a positive GAD antibody test of 101 WHO units or more on two separate occasions.
4. Age 18 +
5. The patient did not start on insulin within 1 month of diagnosis
6. Written informed consent to participate in the study.
7. Ability to comply with all study requirements.

Exclusion Criteria:

1. Pregnant or breast-feeding females and females who plan pregnancy or breast-feeding during the course of the study.
2. A history of:

   Diabetes that is a result of pancreatic injury, or secondary forms of diabetes, e.g., Cushing's syndrome and acromegaly.

   Acute metabolic diabetic complications such as ketoacidosis or hyperosmolar state (coma) within the past 6 months
3. Acute infections, which may affect blood glucose control within 4 weeks prior to visit 1.
4. Malignancy including leukaemia and lymphoma (not including basal cell skin cancer) within the last 5 years.
5. The patient has a known immune deficiency from any disease, or a condition associated with an immune deficiency.
6. The patient is receiving immunosuppressive or immunomodulating agents or cytotoxic therapy, or any medication that, in the opinion of the site investigator, might interfere with the study.
7. Any of the following significant laboratory abnormalities:

   * Patients with severe renal failure as defined previous renal transplant or currently having renal dialysis or GFR <30.
   * Clinically significant laboratory abnormalities, confirmed by repeat measurement, that may interfere with the assessment of safety and/or efficacy of the study drug, other than hyperglycemia and glycosuria at visit 1.
   * Severe ketonuria (+++ on urine sticks testing; ++ on repeated urine sticks testing).
8. The patient is a known or suspected drug abuser.
9. The patient has chronic hepatitis or liver cirrhosis, or any other chronic liver disease.
10. The patient is known to test positive for hepatitis B antigens or hepatitis C antibodies
11. The patient is known to test positive for HIV antibodies.
12. The patient has any significant diseases or conditions, including psychiatric disorders and substance abuse that, in the opinion of the site investigator, are likely to affect the patient's response to treatment or their ability to complete the study.
13. The patient has chronic haematological disease.
14. The patient has had a severe blood loss (>400 mL, e.g., blood donation) within 2 months before the first dosing of the study medication.
15. The patient has known proliferative retinopathy.
16. Patient has had stage 3-4 heart failure.
17. The patient is participating in another research study which may affect the results of this trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Change in fasting serum C-peptide level over 24 months and (2) change in HbA1c level over 24 months in patients with LADA. | 24 months

SECONDARY OUTCOMES:
Hypoglycaemic events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sinead Brophy, Principal Investigator — Swansea University; Stephen Bain, Study Director — Swansea University
Locations (2):
- United Kingdom (2):
  - Diabetes Unit, Cardiff, Wales
  - Clinical Research Unit, Swansea, Wales

REFERENCES:
- [Background] Brophy S, Davies H, Bain S, Stephens JW, Cheung WY, Richards K, Wareham K, Beaverstock C, Lloyd J, Page D, Williams M, Russell I, Williams R. Randomized, controlled, parallel-group prospective study to investigate the clinical effectiveness of early insulin treatment in patients with latent autoimmune diabetes in adults. BMC Endocr Disord. 2008 Jul 24;8:8. doi: 10.1186/1472-6823-8-8. PMID 18652676